CLINICAL TRIAL: NCT05951985
Title: High Intensity Functional Training for Individuals With Neurologic Diagnoses and Their Care Partners: A 2-Year Longitudinal Study
Brief Title: High Intensity Functional Training for Individuals With Neurologic Diagnoses and Their Care Partners
Acronym: SHIFT-AR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Colleges of Health Education (Other)
Responsible Party: Principal Investigator, Reed Handlery, Assistant Professor, Arkansas Colleges of Health Education
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACHE-2023-0114
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Neurologic Disorder; Parkinson Disease; Spinal Cord Injuries; Spina Bifida; Stroke; Poliomyelitis; Multiple Sclerosis; Brain Injuries
Keywords: hift; exercise
MeSH Terms: conditions — Nervous System Diseases; Parkinson Disease; Spinal Cord Injuries; Spinal Dysraphism; Stroke; Poliomyelitis; Multiple Sclerosis; Brain Injuries; Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal with assessments occurring quarterly over the course of two years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIFT Exercise (Experimental): In this single group design, all participants will be provided with up to two years of twice weekly supervised group exercise.
  Interventions: Behavioral: HIFT

INTERVENTIONS:
Behavioral: HIFT — Exercise sessions will be 60 to 75 minutes in duration and be a combination of resistance, aerobic, and balance exercise, with emphasis on functional movements performed at a high intensity. Exercises will be tailored/modified to meet the needs of each participant.

SUMMARY:
Individuals with and without neurologic diagnoses greatly benefit from participation in regular exercise but the majority are physically inactive. This is an issue for both them and their care partners as their health is often linked. This study aims to examine the long-term physical and psychosocial effects of structured, group-based, high intensity functional training (HIFT) exercise for people with neurologic diagnoses and their care partners.

DETAILED DESCRIPTION:
Over the course of two years, this study will provide no-cost, twice weekly, group-based, HIFT exercise for people with neurologic diagnoses and their care partners. All participants will be required to have physician or advanced practice provider clearance to exercise. All participants will be evaluated by a physical therapist at no-cost prior to beginning the intervention to assess eligibility for the study. All eligible participants will complete a demographics questionnaire, questionnaires regarding physical and psychosocial health, and a battery of physical tests assessing mobility, strength, endurance, and balance. Participants' physical activity levels will also be monitored throughout the study through accelerometers.

Participants will participate in a maximum of twice weekly HIFT exercise for up to 2 years. All exercise programming will be led by licensed physical therapists with assistance from Doctor of Physical Therapy students. All exercise staff will be Cardiopulmonary resuscitation/basic life support certified and an automated external defibrillator will be available onsite. Exercise classes will utilize HIFT, which includes various exercises that are functional and to be performed at a high intensity. Exercises will include aerobic, resistance, and/or balance training and align with the 2018 Physical Activity Guidelines for Americans.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age
* Participants must be able to communicate and read in English
* Participants must have physician and/or advanced practice provider clearance to exercise
* Participants must have a neurologic diagnosis (e.g., spinal cord injury, Parkinson's, brain injury, stroke, poliomyelitis, multiple sclerosis, spina bifida, etc.) OR participants must be care partner of a person with neurologic diagnosis.
* Participants must possess at least 4/5 elbow flexion strength bilaterally
* Participants must be able to locomote independently (i.e., ambulate or propel a manual or power wheelchair independently).
* Participants must provide their own transportation to/from the research study

Exclusion Criteria:

* Participants will be excluded if they fail to meet any of the inclusion requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Participant Attendance at 24 months | After 24 months of intervention
  The percentage of intervention sessions attended by participants.

SECONDARY OUTCOMES:
Change in lower extremity functional strength at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Lower extremity strength will be measured via functional test (Five Times Sit to Stand). This test records the amount of time taken to rise and sit to and from a chair five consecutive times. Faster times indicate greater lower extremity strength.
hange in Parkinson's Disease Questionnaire - 39 (PDQ-39) at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The PDQ-39 is a 39-item participant-reported questionnaire which assesses health-related quality of life across 8 domains (mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, bodily discomfort). Participants respond to each item using a 5-point Likert scale from 0 (never) to 4 (always). Items in each domain are scored by expressing summed item scores as a percentage (ranging from 0 to 100%). Lower scores indicate better quality of life.
Change in fast-paced gait speed at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Fast-paced walking speed will be measured via 10 meter walk test, which has individuals walk 10 meters with the middle 6 meters timed; two trials are performed and the average time is taken. Faster walking speeds indicate greater mobility with walking.
Change in fast-paced wheelchair propulsion speed at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Fast-paced propulsion speed will be measured via wheelchair propulsion test, which has individuals propel 10 meters and are timed; two trials are performed and the average time is taken. Faster propulsion speeds indicate greater mobility with wheelchair propulsion.
Change in 6 Minute Walk Test at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The 6 Minute Walk Test measures a participants ability to cover as much distance (measured in meters) as possible while walking for 6 minutes. Participants will walk along a pre-defined pathway for 6 minutes, resting as needed. The test is a measure of walking endurance with further distances indicating greater endurance.
Change in 6 Minute Propulsion Test at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The 6 Minute Propulsion Test measures a participants ability to cover as much distance (measured in meters) as possible while propelling a wheelchair for 6 minutes. The test is a measure of aerobic endurance with further distances indicating greater endurance.
Change in Movement Disorder Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The MDS-UPDRS measures disability as a result of Parkinson's and allows tracking for progression of the disease. The scale has four parts (1, mentation, behavior and mood, 2, activities of daily living, 3, motor examination, and 4, complications of therapy. Each parkinsonian sign or symptom is ranked on a 5-point Likert scale (ranging from 0 to 4) with higher scores indicating greater impairments. The minimum score on the entire scale is 0 and the maximum is 199.
Change in accelerometer-measured moderate-to-vigorous physical activity at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Physical activity levels will be measured via thigh or wrist-worn accelerometer (activPAL or ActiGraph). These small devices will be worn on the less affected thigh or wrist (or non-dominant thigh or wrist for care partners). Through collecting acceleration data, different intensities of physical activity will be inferred (i.e light, moderate and vigorous intensity physical activity), with moderate-to-vigorous intensity physical activity being used as the primary outcome measure. At all time points, participants will wear the accelerometer for 7 consecutive days.
Participant Retention at 24 months | After 24 months of intervention
  The number and percentage of participants who remain in the study through the final measurement point at 24 months.
Participant Recruitment Rates | Throughout the 24 months study period
  The number of participants recruited will be reported as a percentage of total participants contacted for study participation.
Change in four square step test at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The four square step test measures stepping balance as the time taken to step clockwise and counterclockwise in a square pattern. Faster times indicate greater balance.
YMCA Bench Press Test at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The YMCA Bench Press Test measures muscular endurance of the upper body. The test requires participants to complete as many repetitions of barbell bench press as they can with good form. Greater number of repetitions indicates greater muscular endurance.
30 second peak power test at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  The 30 second peak power test measures anaerobic power produced (in watts) over 30 seconds on a ski ergometer. Greater wattage indicates greater anaerobic power.
Change in self-reported exercise confidence at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Change will be reported using a visual analogue scale where participants rate their confidence from not confident at all to completely confident.
Change in self-reported pain at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Change will be reported using a visual analogue scale where participants rate their pain from no pain to worst possible pain.
Change in self-reported sleep quality at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Change will be reported using a visual analogue scale where participants rate their sleep quality from poor to exceptional.
Change in self-reported social support at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Change will be reported using a visual analogue scale where participants rate their level of social support from people in the intervention and those outside the intervention. The scale goes from poor to exceptional social support.
Change in self-reported physical ability at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Change will be reported using a visual analogue scale where participants rate their level of ability from poor to exceptional on attributes of mobility, power, endurance/stamina, strength and balance.
Self-reported safety with program at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Using a visual analogue scale, participants rate their feelings of safety with the intervention at 24 months. Scores range from not safe at all to exceptionally safe.
Self-reported satisfaction with coach supervision at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Using a visual analogue scale, participants rate their feelings of satisfaction with coach supervision during the intervention at 24 months. Scores range from not satisfied at all to extremely satisfied.
Self-reported feelings of inclusion at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Using a visual analogue scale, participants rate their feelings of inclusion during the intervention at 24 months. Scores range from minimally included to maximally included.
Self-reported feelings of exercise intensity at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Using a visual analogue scale, participants rate their feelings of exercise intensity during the intervention at 24 months. Scores range from low intensity to high intensity exercise.
Self-reported feelings of exercise variety at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Using a visual analogue scale, participants rate their feelings on exercise variety during the intervention at 24 months. Scores range from low exercise variety to high exercise variety.
Self-reported feelings of exercise applicability in real life at 24 months | After, 3, 6, 9, 12, 15, 18, 21 and 24 months of intervention
  Using a visual analogue scale, participants rate their feelings on applicability of exercises to real life during the intervention at 24 months. Scores range from not applicable at all to extremely applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Colleges of Health Education, Fort Smith, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided
All non-identifiable data may be made available to other researchers upon request.

REFERENCES:
- [Background] Schenkman M, Moore CG, Kohrt WM, Hall DA, Delitto A, Comella CL, Josbeno DA, Christiansen CL, Berman BD, Kluger BM, Melanson EL, Jain S, Robichaud JA, Poon C, Corcos DM. Effect of High-Intensity Treadmill Exercise on Motor Symptoms in Patients With De Novo Parkinson Disease: A Phase 2 Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):219-226. doi: 10.1001/jamaneurol.2017.3517. PMID 29228079
- [Background] Ellis TD, Cavanaugh JT, DeAngelis T, Hendron K, Thomas CA, Saint-Hilaire M, Pencina K, Latham NK. Comparative Effectiveness of mHealth-Supported Exercise Compared With Exercise Alone for People With Parkinson Disease: Randomized Controlled Pilot Study. Phys Ther. 2019 Feb 1;99(2):203-216. doi: 10.1093/ptj/pzy131. PMID 30715489
- [Background] Feito Y, Heinrich KM, Butcher SJ, Poston WSC. High-Intensity Functional Training (HIFT): Definition and Research Implications for Improved Fitness. Sports (Basel). 2018 Aug 7;6(3):76. doi: 10.3390/sports6030076. PMID 30087252
- [Background] Adams J, Lai B, Rimmer J, Powell D, Yarar-Fisher C, Oster RA, Fisher G. Telehealth high-intensity interval exercise and cardiometabolic health in spinal cord injury. Trials. 2022 Aug 4;23(1):633. doi: 10.1186/s13063-022-06585-2. PMID 35927708